CLINICAL TRIAL: NCT06974240
Title: Social Robotics Intervention for Improving Socio-Pragmatic Skills in Autism: A Randomized Controlled Trial
Brief Title: Social Robotics for Autism
Acronym: SRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Collaborators: Messina, Italy (Other)
Responsible Party: Principal Investigator, Flavia Marino, Head of Unit, Istituto per la Ricerca e l'Innovazione Biomedica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNR-IRIB-PRO-2025-003
Record Dates: First submitted 2025-04-24; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: autism; social robot; social pragmatic skills; intervention; social skills; educational technologies
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Social Skills | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group with social robot (Experimental): Ten children with ASD, aged between 8 and 13 years and with verbal IQs above 75, will be included in the trial following an assessment of their socio-pragmatic skills. They will be randomly assigned to either the control group or the experimental group. Participants in the experimental group will undergo an intervention aimed at developing and/or enhancing socio-pragmatic skills through the mediation of a social robot.
  Interventions: Other: Experimental Group
- Control Group (Other): Ten children with ASD, aged between 8 and 13 years and with verbal IQs above 75, will be included in the trial following an assessment of their socio-pragmatic skills. Children in the control group will follow the same protocol of Experimental Group delivered through a therapist-led group format.
  Interventions: Other: control group

INTERVENTIONS:
Other: Experimental Group — The training sessions were carried out following a strict order. The first phase was dedicated to improving group social skills. The beginning of the session was dedicated to greetings between participants and questions of social interest. During the second phase, videos were shown and participants answered targeted questions asked by the Nao Robot to understand if the child had correctly interpreted the general meaning of the story and to determine the degree of awareness that the expression should be understood in a non-literal sense. In the third phase, a role play was performed among the participants, which re-enacted the situations seen in the videos, involving all the members of the group in turn. During the last phase, participants were asked to share experiences in their lives in which they had used or could have used the pragmatic skill just analyzed. The protocol included 15 phases over 31 sessions, each lasting 45 minutes, twice a week.
  Arms: Experimental Group with social robot
Other: control group — The entire intervention was carried out in a group entirely mediated by an operator without the use of a social robot. The first phase is dedicated to improving group social skills. The beginning of the session was dedicated to greetings between participants and questions of social interest. During the second phase, stories were read and participants answered target questions to understand if the child had correctly interpreted the general meaning of the story and to determine the degree of awareness that the expression should be understood in a non-literal sense. In the third phase, a role play was performed among the participants, in which all members of the group participated in turn, recalling the situations seen in the videos. During the last phase, participants were asked to share experiences from their lives in which they used or could use the pragmatic skill just analyzed. The protocol included 15 phases over 31 sessions, each lasting 45 minutes, twice a week.
  Arms: Control Group

SUMMARY:
Socio-pragmatics focuses on the study of language in the context of social interactions. It explores how individuals use language to communicate effectively in specific social situations, taking into consideration the social, cultural and contextual factors that influence communication. Socio-pragmatics analyzes linguistic and nonlinguistic behaviors, such as gestures, facial expressions, tone of voice, and posture, to understand intended meaning, social implications, and shared communicative norms. Children with autism often present difficulties in social-pragmatic skills.

The integration of advanced technologies can play a crucial role in innovative approaches to the development of this skill.

In this experimental protocol, an attempt will be made to demonstrate the effectiveness of training through the use of social robots by comparing the performance of an ASD group performing a treatment using social robots with a control group performing the same in a traditional manner.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 8 and 13 years
* Clinical diagnosis of ASD according to DSM-5 criteria by a licensed child neuropsychiatrist
* Verbal and performance IQ > 75 and total IQ > 85, assessed with the WISC-IV
* No current aggressive behavior or severe oppositional tendencies
* No hearing, vision, or physical impairments that could interfere with participation
* Not currently taking any psychotropic medications

Exclusion Criteria:

* Absence of a clinical diagnosis of ASD based on DSM-5 criteria
* Verbal or performance IQ ≤ 75, or total IQ ≤ 85 as assessed by WISC-IV
* Presence of aggressive behavior or severe oppositional tendencies
* Hearing, vision, or physical impairments that could hinder participation in the intervention
* Current use of psychotropic medications

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Wechsler Intelligence Scale for Children 4° edizione (WISC-IV) | Baseline assessment at Day 1 (prior to intervention); the test requires approximately 56-80 minutes to complete.
  Wechsler Intelligence Scale for Children 4° edizione (WISC-IV) is a clinical tool for assessing the cognitive abilities of children and young people between the ages of 6 years and 16 years and 11 months.
Language Pragmatic Abilities (APL) -MEDEA | Baseline assessment at Day 1 (pre-intervention) and post-intervention assessment at 3 months (at the end of the intervention); each test session lasts approximately 30-45 minutes.
  The APL MEDEA is a standardized assessment tool specifically designed to evaluate socio-pragmatic skills in individuals aged 5 to 14 years. This test measures various aspects of pragmatic language skills that are essential for effective communication within social contexts.
  The main objective of the APL MEDEA is to assess pragmatic language skills employed during everyday interactions, including the understanding and appropriate use of language in various social situations, recognition of social cues, and effective conversational strategies. The total score ranges from 0 to 68.

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Marino, Principal Investigator — Italy Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR)
Locations (1):
- Italy Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR), Messina, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holeva V, Nikopoulou VA, Lytridis C, Bazinas C, Kechayas P, Sidiropoulos G, Papadopoulou M, Kerasidou MD, Karatsioras C, Geronikola N, Papakostas GA, Kaburlasos VG, Evangeliou A. Effectiveness of a Robot-Assisted Psychological Intervention for Children with Autism Spectrum Disorder. J Autism Dev Disord. 2024 Feb;54(2):577-593. doi: 10.1007/s10803-022-05796-5. Epub 2022 Nov 4. PMID 36331688
- [Background] Taheri, A., Shariati, A., Heidari, R., Shahab, M., Alemi, M., & Meghdari, A. (2021). Impacts of using a social robot to teach music to children with low-functioning autism. Paladyn, Journal of Behavioral Robotics, 12(1), 256-275.
- [Background] So WC, Cheng CH, Law WW, Wong T, Lee C, Kwok FY, Lee SH, Lam KY. Robot dramas may improve joint attention of Chinese-speaking low-functioning children with autism: stepped wedge trials. Disabil Rehabil Assist Technol. 2023 Feb;18(2):195-204. doi: 10.1080/17483107.2020.1841836. Epub 2020 Nov 13. PMID 33186058